CLINICAL TRIAL: NCT05952323
Title: Comparison of Different Teaching Methods in Increasing Nursing Students' Competencies for Safe Use of Medical Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha CENGİZ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2023/4644
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Nurse's Role
Keywords: Competency; Medical devices; Nursing; Teach-Back; Students; Video-assisted teaching

STUDY DESIGN:
Intervention Model Description: A two-tailed test at a 5% significance level with a power of 95% indicated that a sample size of 90 was required for an effect size of 0.37. Considering potential data loss during the research process, 5 students will included in each group (teach-back group = 35, video-assisted teaching group = 35, control group = 35). Since it is anticipated that student performance may affect competency, students will be stratified based on their overall academic average in this study. Subsequently, computer-assisted randomization will be used to assign an equal number of students from each stratum to each group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): After obtaining the necessary legal and ethical permissions for data collection, the research will commence. During this stage of the study, participants who agree to take part in the research will be asked to fill out the informed consent form. To obtain the pre-test data for the research, all forms will be filled out.
  Students receiving standard care and continuing practice will be provided with information about the research. Pre-test and post-test data from the control group will be obtained concurrently with the study groups.
- Teach-back group (Experimental): To obtain the pre-test data for the research, all forms will be filled out. According to the prepared educational materials for medical devices, students will be trained using the teach-back method. After the training, students will be asked to demonstrate their skills in using medical devices then two weeks after the pre-test. The researcher will use the Medical Device Usage Competency Observer Evaluation Form to assess the student's competency in using medical devices and Medical Device Usage Competency Knowledge Test and the Medical Device Usage Competency Self-Assessment Form for post-test data.
  Interventions: Other: Teach-back
- Video-assisted teaching group (Experimental): After obtaining the pre-test data, students will be sent educational videos related to medical devices and asked to watch them. Then two weeks after sending the videos, students will be requested to demonstrate their skills in using medical devices. The researcher will assess the students' medical device usage competencies using the Medical Device Usage Competency Observer Evaluation Form, Medical Device Usage Competency Knowledge Test, and the Medical Device Usage Competency Self-Assessment Form for post-test data.
  Interventions: Other: Video-assisted teaching

INTERVENTIONS:
Other: Teach-back — According to the prepared educational materials for medical devices, students will be trained using the teach-back method.
  Arms: Teach-back group
Other: Video-assisted teaching — Students will be sent educational videos related to medical devices and asked to watch them.
  Arms: Video-assisted teaching group

SUMMARY:
A significant portion of nursing practice involves the application of technical skills and the use of medical devices. Nowadays, the number and complexity of medical devices in healthcare settings are increasing. Therefore, it is of great importance for nurses to have appropriate knowledge and skills in this field to provide adequate and safe patient care.

DETAILED DESCRIPTION:
Nursing education plays a vital role in equipping student nurses with the necessary knowledge and skills to become competent and reliable healthcare professionals. The use of interactive methods in education has a significant impact on enhancing nursing students' competencies. There is a lack of sufficient research in the literature regarding the effectiveness of teach-back and video-supported instruction on the safe use of medical devices. Hence, this study aims to compare the effectiveness of teach-back and video-supported teaching methods in enhancing nursing students' competencies in the safe use of medical devices.

The research will be conducted between September 2023 and May 2024 in a designated training room at the hospital where the clinical training of senior nursing students takes place. The sample of the study will consist of a total of 105 students, who will be divided into three groups using randomization: a teach-back group (35 students), a video-supported instruction group (35 students), and a control group (35 students). Data will be collected using the Student Information Form, Medical Device Usage Competency Self-Assessment Form, Medical Device Usage Competency Knowledge Test, and Medical Device Usage Competency Observer Evaluation Form. For data analysis, the normality of the data will first be determined using the Shapiro-Wilk normality test. Parametric tests will be used for normally distributed data, while non-parametric tests will be used for non-normally distributed data.

ELIGIBILITY:
Inclusion Criteria:

* Be a senior nursing student
* Be taking the Nursing Care Management course for the first time
* Have no previous work experience as a nurse outside of clinical training
* Have no visual, auditory, cognitive, or perceptual impairments
* Not have received any planned training program or course specifically on the use of infusion pumps, patient monitors, and suction devices
* Have access to an Android phone or computer for the study.

Exclusion Criteria:

* Have graduated from a Health Vocational High School.
* Be taking the Nursing Care Management course for the second time.
* Obtain a score above the predetermined threshold on the knowledge test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
The Medical Device Usage Competency Self-Assessment Form | 6 months
  The Medical Device Usage Competency Self-Assessment Form is a tool used to assess an individual's self-perceived competency in using medical devices. It typically consists of a series of questions or statements related to different aspects of medical device usage, such as knowledge, skills, and confidence. A research form has been developed by the researcher through a literature review. The content validity of the form will be determined and Cronbach's Alpha coefficient will be examined. The form is designed using a five-point Likert scale to capture participants' opinions on medical device usage competency.
The Medical Device Usage Competency Knowledge Test | 6 months
  It typically consists of a series of questions or scenarios related to different aspects of medical devices, including their purpose, indications, proper usage techniques, safety precautions, troubleshooting, and maintenance. The test aims to evaluate the individual's factual knowledge and comprehension of essential information related to medical device usage. Knowledge Test has been developed by the researcher based on the literature review. Expert opinions will be sought to validate the content of the test. The test will consist of multiple-choice and true/false questions.
The Medical Device Usage Competency Observer Evaluation Form | 6 months
  It is typically completed by trained observers or evaluators who assess the individual's performance in using medical devices based on specific criteria. The form serves as a standardized assessment tool to gather objective data on the individual's practical skills and abilities in handling medical devices. The form has been developed by the researcher based on the available literature. The content validity of the steps in the form will be determined based on expert opinions.

CONTACTS AND LOCATIONS:
Locations (1):
- Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This research is a doctoral thesis study. The research is expected to be completed.